CLINICAL TRIAL: NCT01417481
Title: Evaluation of the Capability of a Glycine Oral Supplement for Diminishing Bronchial Inflammation in Children With Cystic Fibrosis
Brief Title: Effect of Glycine in Cystic Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Some of the researchers finished their participation in the study.
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other); Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Mario H. Vargas, Senior Researcher, Instituto Nacional de Enfermedades Respiratorias
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Glycine in CF
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; glycine; airway inflammation
MeSH Terms: conditions — Cystic Fibrosis | interventions — Glycine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glycine (Active Comparator): Patients will receive a daily oral supplement of 0.5 g/kg glycine dissolved in water.
  Interventions: Dietary Supplement: Glycine
- Placebo (Placebo Comparator): Patients will receive a daily supplement of 0.5 g/kg sugar glass dissolved in water.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Glycine — Daily oral supplement of glycine at a dose of 0.5 g/kg divided in three doses during 8 weeks
  Other Names: aminoacetic acid
  Arms: Glycine
Dietary Supplement: Placebo — Daily oral administration of placebo (sugar glass) at a dose of 0.5 g/kg divided in three doses during 8 weeks
  Other Names: sugar glass
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate if glycine, orally administered in a daily dose of 0.5 g/kg during 8 weeks, can ameliorate the airway inflammation in children with cystic fibrosis, as compared with placebo. During all of the study children will receive their usual treatment for cystic fibrosis.

DETAILED DESCRIPTION:
Background. Cystic fibrosis (CF) is a genetic disorder caused by a mutation in a gene that codifies for a chloride channel named "cystic fibrosis transmembrane regulator" (CFTR). In the lungs this results in thick and dehydrated mucus that tends to cause obstruction of the bronchial lumen. Neutrophils and proinflammatory substances have been detected in bronchoalveolar lavage fluid of children with CF who have no bacterial infection. This inflammation conditions a vicious circle in which airways are colonized by bacteria that further increase inflammation. Persistent inflammation leads to irreversible changes in airways, which become distorted. Therefore, a key step in CF treatment is reduction of airway inflammation, for which long-term use of corticosteroids, ibuprofen or macrolides may be indicated.

Glycine and its antiinflammatory effect. Glycine is the most simple aminoacid, but it is also an agonist of the glycine receptors (GlyR) that, when activated, cause that cells such as Kupffer cells, alveolar macrophages and neutrophils decrease their sensitivity to proinflammatory agents. Orally administered glycine has been used for some illnesses, and it has been noticed that it is well tolerated. Considering that children with CF have an intense inflammatory process in the airways, here we propose to use glycine as antiinflammatory agent.

Problem statement. Can a glycine oral supplement decrease the airway inflammation in children with CF?

Hypothesis. Compared with placebo, a daily supplement of glycine administered for 8 weeks to children with CF produce a statistically significant decrease of bronchial inflammation, measured by the concentration of neutrophils and inflammatory substances in sputum and peripheral blood, as well as by respiratory symptoms and spirometry.

Main objective: To determine whether a daily supplement of 0.5 g/kg glycine for 8 weeks significantly decrease the concentration, including neutrophils, interleukin(IL)-1β, IL-6, IL-8, tumor necrosis factor alpha (TNF-α), and myeloperoxidase, in sputum and peripheral blood of children with CF.

Secondary Objectives:

1. To determine if glycine can improve respiratory symptoms, including decreased amount and better fluidity of sputum.
2. To determine if glycine can improve spirometric variables.

Study design. This will be a randomized, placebo controlled, blinded, two-arms, cross-over clinical trial. Patients will receive glycine or placebo during the initial 8 weeks (initial phase), and after a 2 weeks washout period, they will receive the alternate treatment during another 8 weeks (second phase).

Material and methods: Children with CF fulfilling the selection criteria will be studied if their parents accept their participation. They will be randomly assigned to one of two groups. The experimental group will receive glycine and the control group will receive placebo (sugar glass), both at doses of 0.5 g/kg divided in 3 doses per os dissolved in any liquid. At study entry and at weeks 4, 8, 10, 14 and 18 we will collect a 2 ml blood sample and a sputum sample, and the children will be submitted to spirometry. A daily symptom questionnaire will be filled by the parents.

Statistical analysis: Each variable will be compared between experimental and control groups using Student's t test (or Mann Whitney U test if lacking normal distribution). Sample size: There are no previous studies that allow us to calculate a sample size. For convenience, it is estimated that 30 children can be included.

Time to complete: 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex
* Between 5 and 15 years of age
* With CF diagnosed according to established criteria
* Without changes in the CF treatment in the last 30 days
* Without CF exacerbation in the last 30 days
* Without acute respiratory infection (e.g., common cold) in the last 15 days
* Informed consent letter signed by their parents or legal guardians

Exclusion Criteria:

* Children with CF that had participated in a research protocol in the last 3 months
* Presence of serious adverse effects attributable to glycine, in which case the result will be considered as therapeutic failure in the statistical analysis
* Development of a CF exacerbation, in which case the available data so far collected will be included in the statistical analysis

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario H Vargas, MD, MSc, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (3):
- Mexico (3):
  - Hospital Infantil de México, Mexico City
  - Unidad de Investigación Médica en Enfermedades Respiratorias, Hospital de Pediatría, CMN SXXI, IMSS, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias, Mexico City

REFERENCES:
- [Background] Cohen-Cymberknoh M, Shoseyov D, Kerem E. Managing cystic fibrosis: strategies that increase life expectancy and improve quality of life. Am J Respir Crit Care Med. 2011 Jun 1;183(11):1463-71. doi: 10.1164/rccm.201009-1478CI. Epub 2011 Feb 17. PMID 21330455
- [Background] Wheeler MD, Ikejema K, Enomoto N, Stacklewitz RF, Seabra V, Zhong Z, Yin M, Schemmer P, Rose ML, Rusyn I, Bradford B, Thurman RG. Glycine: a new anti-inflammatory immunonutrient. Cell Mol Life Sci. 1999 Nov 30;56(9-10):843-56. doi: 10.1007/s000180050030. PMID 11212343
- [Background] Wheeler MD, Rose ML, Yamashima S, Enomoto N, Seabra V, Madren J, Thurman RG. Dietary glycine blunts lung inflammatory cell influx following acute endotoxin. Am J Physiol Lung Cell Mol Physiol. 2000 Aug;279(2):L390-8. doi: 10.1152/ajplung.2000.279.2.L390. PMID 10926563
- [Background] Garcia-Macedo R, Sanchez-Munoz F, Almanza-Perez JC, Duran-Reyes G, Alarcon-Aguilar F, Cruz M. Glycine increases mRNA adiponectin and diminishes pro-inflammatory adipokines expression in 3T3-L1 cells. Eur J Pharmacol. 2008 Jun 10;587(1-3):317-21. doi: 10.1016/j.ejphar.2008.03.051. Epub 2008 Apr 8. PMID 18499099
- [Derived] Vargas MH, Del-Razo-Rodriguez R, Lopez-Garcia A, Lezana-Fernandez JL, Chavez J, Furuya MEY, Marin-Santana JC. Effect of oral glycine on the clinical, spirometric and inflammatory status in subjects with cystic fibrosis: a pilot randomized trial. BMC Pulm Med. 2017 Dec 15;17(1):206. doi: 10.1186/s12890-017-0528-x. PMID 29246256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients attending the Hospital Infantil de México and the Instituto Mexicano del Seguro Social (both in Mexico city) were recruited from March 7, 2012 to October 31, 2012. The two arms of the study were: 1) Glycine, then placebo, and 2) Placebo, then glycine.
Groups:
- Glycine, Then Placebo: First intervention (8 weeks) with Glycine (0.5 g/kg/day divided in three doses).
  Washout period of 2 weeks. Second intervention (8 weeks) with Placebo (sugar glass, 0.5 g/kg/day divided in three doses).
- Placebo, Then Glycine: First intervention (8 weeks) with Placebo (sugar glass, 0.5 g/kg/day divided in three doses).
  Washout period of 2 weeks. Second intervention (8 weeks) with Glycine (0.5 g/kg/day divided in three doses).
Period: First Intervention (8 Weeks)
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine
Started | 8 | 7
Completed | 8 | 5
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Washout (2 Weeks)
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine
Started | 8 | 5
Completed | 8 | 5
Not Completed | 0 | 0
Period: Second Period (8 Weeks)
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine
Started | 8 | 5
Completed | 8 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The total number of patiens was fewer than planned mainly because other protocols were running concurrently. The protocolo had to be concluded because some of the researchers finished their participation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycine, Then Placebo | Placebo, Then Glycine | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants] — During the course of the study, inclusion criteria was expanded to include subjects older than 15 years of age.
  Participants
    <=18 years | 6 | 7 | 13
    Between 18 and 65 years | 2 | 0 | 2
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.39 (5.82) | 11.00 (4.01) | 12.81 (5.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  Mexico | 8 | 7 | 15

OUTCOME MEASURES:

1. Secondary Outcome: Changes in Clinical Data Scores (Other Than Sputum Production, Dyspnea and Global Symptoms)
Description: To correct for the baseline variability, all measurements were expressed as percentage of baseline (value at week 8 with respect to baseline value [beginning of the glycine or placebo period, respectively]).
  Each respiratory symptom (Cough severity, Sputum features, Appetite, Dyspnea, and Energy perception) was evaluated in a 5-options Likert scale, ranging from 1 (better) to 5 (worse). The total score was computed by the simple sum of the five symptoms.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: Percentage of baseline
Groups:
- Glycine: All study participants receiving a daily oral supplement of 0.5 g/kg glycine dissolved in water during 8 weeks.
- Placebo: All study participants receiving a daily oral supplement of 0.5 g/kg placebo (sugar glass) dissolved in water during 8 weeks.
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of baseline
  Cough questionnaire score | 81.1 (12.6) | 89.1 (4.9)
  Appetite questionnaire score | 89.1 (11.0) | 132.1 (25.4)
  Energy questionnaire score | 84.6 (7.4) | 111.5 (16.2)
  Body weight | 101.6 (1.1) | 103.6 (1.0)
  Height | 100.5 (0.2) | 100.5 (0.2)
  Heart rate | 103.5 (6.0) | 98.1 (3.0)
  Respiratory rate | 94.8 (5.5) | 109.0 (6.4)
  Temperature | 100.0 (0.3) | 100.1 (0.5)
Statistical Analysis 1: Comparison: Glycine vs Placebo; Test type: Superiority or Other; p > 0.05, t-test, 1 sided; Due to the cross-over, a paired analysis was done. The hypothesis was that glycine will improve variables, and thus significance was set at one-tail

2. Primary Outcome: Changes in Serum Concentration of Inflammatory Biomarkers (Other Than TNF-alpha)
Description: To correct for the baseline variability, all measurements were expressed as percentage of baseline (value at week 8 with respect to baseline value [beginning of the glycine or placebo period, respectively]). Then, percentages were log-transformed to adjust to a normal distribution.
Time Frame: 8 weeks
Population: From the 13 patients who initiated the study, some parents did not give consent for blood sampling, and some children refused the venous puncture at some visits. Thus, only a non-paired population of 9 children per group could be analyzed.
Measure: Mean (Standard Error); unit: log (percent change)
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 9 | 9
log (percent change)
  Myeloperoxidase | -0.4361 (0.2184) | -0.2906 (0.2877)
  IL-1 | -0.1635 (0.1467) | -0.0352 (0.1294)
  IL-4 | 0.2964 (0.1420) | 0.1470 (0.2223)
  IL-6 | 0.0085 (0.2064) | 0.2255 (0.1865)
  IL-7 | 0.0356 (0.0613) | 0.0819 (0.0986)
  IL-8 | -0.1466 (0.2981) | -0.2364 (0.1761)
  IL-12 | 0.3203 (0.1449) | 0.2603 (0.2117)
  IL-13 | -0.0561 (0.1684) | 0.1953 (0.1849)
  G-CSF | -0.0776 (0.1554) | 0.2272 (0.1983)
  IFN-gamma | 0.3272 (0.1761) | 0.3639 (0.2505)
  MCP-1 | -0.0836 (0.1041) | 0.0472 (0.0894)
  MIP-1beta | 0.0330 (0.1426) | -0.0608 (0.0963)
Statistical Analysis 1: Comparison: Glycine vs Placebo; Test type: Superiority or Other; p > 0.05, t-test, 1 sided; The hypothesis was that glycine will improve inflammatory biomarkers, and thus statistical significance was set at one-tail

3. Primary Outcome: Changes in Sputum Concentration of Inflammatory Biomarkers (Other Than IL-6 and G-CSF)
Description: To correct for the baseline variability, all measurements were expressed as percentage of baseline (value at week 8 with respect to baseline value [beginning of the glycine or placebo period, respectively]). Then, percentage change was log-transformed to adjust to a normal distribution.
Time Frame: 8 weeks
Population: From the 13 patients who initiated the study, some children at some visits could not give an appropriate sputum sample. Thus, only a non-paired population of 9 (glycine group) and 11 (placebo group) children could be analyzed.
Measure: Mean (Standard Error); unit: log (percent change)
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 9 | 11
log (percent change)
  Myeloperoxidase | 0.1294 (0.2204) | 0.0669 (0.1725)
  IL-1 | -0.0918 (0.1552) | -0.0102 (0.1329)
  IL-2 | 0.0233 (0.0828) | -0.0274 (0.1243)
  IL-4 | -0.0161 (0.0482) | 0.0522 (0.0671)
  IL-5 | 0.2498 (0.1855) | 0.1304 (0.1864)
  IL-7 | 0.0611 (0.0852) | 0.1387 (0.1028)
  IL-8 | -0.0824 (0.2311) | 0.0542 (0.0934)
  IL-10 | 0.0549 (0.0847) | 0.0074 (0.0849)
  IL-12 | 0.1675 (0.1443) | 0.0677 (0.1250)
  IL-13 | 0.1630 (0.1379) | 0.0953 (0.1049)
  IL-17 | 0.0680 (0.0411) | 0.1140 (0.0823)
  IFN-gamma | 0.0248 (0.0652) | 0.0649 (0.0730)
  MCP-1 | 0.0042 (0.0694) | 0.2608 (0.2025)
  MIP-1beta | -0.0303 (0.1234) | 0.0977 (0.1207)
  TNF-alpha | 0.0412 (0.1091) | 0.1568 (0.1393)
  GM-CSF | -0.0538 (0.0338) | -0.0822 (0.0468)
Statistical Analysis 1: Comparison: Glycine vs Placebo; Test type: Superiority or Other; p > 0.05, t-test, 1 sided; [statistical method as in outcome 2, analysis 1]

4. Primary Outcome: Changes in Serum Concentration of Inflammatory Biomarkers (TNF-alpha)
Description: as for outcome 2
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log (percent change)
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 9 | 9
log (percent change) | -0.3908 (0.2744) | 0.2035 (0.2384)
Statistical Analysis 1: Comparison: Glycine vs Placebo; Test type: Superiority or Other; p = 0.061, t-test, 1 sided; [statistical method as in outcome 2, analysis 1]

5. Primary Outcome: Changes in Sputum Concentration of Inflammatory Biomarkers (IL-6)
Description: as for outcome 3
Time Frame: 8 weeks
Population: From the 13 patients who initiated the study, some children did not expectorate at some visits. Thus, only a non-paired population of 9 children under glycine and 11 under placebo could be analyzed.
Measure: Mean (Standard Error); unit: log (percent change)
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 9 | 11
log (percent change) | -0.00007 (0.0677) | 0.1739 (0.0838)
Statistical Analysis 1: Comparison: Glycine vs Placebo; Test type: Superiority or Other; p = 0.068, t-test, 1 sided; [statistical method as in outcome 2, analysis 1]

6. Primary Outcome: Changes in Sputum Concentration of Inflammatory Biomarkers (G-CSF)
Description: as for outcome 3
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: log (percent change)
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 9 | 11
log (percent change) | -0.0819 (0.0790) | 0.1668 (0.1022)
Statistical Analysis 1: Comparison: Glycine vs Placebo; Test type: Superiority or Other; p = 0.040, t-test, 1 sided; [statistical method as in outcome 2, analysis 1]

7. Secondary Outcome: Changes in Score for Sputum Production, Dyspnea and Global Symptoms
Description: To correct for the baseline variability, all measurements were expressed as percentage of baseline (value at week 8 with respect to baseline value [beginning of the glycine or placebo period, respectively]).
  In the symptoms questionnaire, each respiratory symptom (Cough severity, Sputum features, Appetite, Dyspnea, and Energy perception) was evaluated in a 5-options Likert scale, ranging from 1 (better) to 5 (worse). The total score was computed by the simple sum of the five symptoms.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: Percentage of baseline
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of baseline
  Sputum questionnaire score | 82.0 (7.0) | 102.6 (10.1)
  Dyspnea questionnaire score | 75.6 (7.5) | 103.8 (10.7)
  Total questionnaire score | 77.7 (5.2) | 98.7 (8.4)
Statistical Analysis 1: Comparison: Glycine vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 1 sided; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Changes in Pulse Oximetry, FEV1/FVC, and FEF50.
Description: To correct for the baseline variability, all measurements were expressed as percentage of baseline (value at week 8 with respect to baseline value [beginning of the glycine or placebo period, respectively]).
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: Percentage of baseline
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of baseline
  Peripheral oxygen saturation (SpO2) | 105.2 (2.5) | 98.9 (1.4)
  FEV1/FVC | 105.2 (2.9) | 94.9 (4.2)
  Forced expiratory flow at 50%FVC (FEF50) | 115.5 (10.4) | 93.1 (7.8)
Statistical Analysis 1: Comparison: Glycine vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 1 sided; Due to the cross-over, paired analysis was done. The hypothesis was that glycine will improve variables, thus significance was set at one-tail

9. Secondary Outcome: Changes in FEV1, FEF25, and FEFmax
Description: as for outcome 8
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: Percentage of baseline
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of baseline
  Forced expiratory volume at first second (FEV1) | 109.7 (6.4) | 91.4 (4.1)
  Forced expiratory flow at 25%FVC (FEF25) | 133.9 (13.6) | 83.3 (7.7)
  Maximal forced expiratory flow (FEFmax, PEFR) | 115.3 (6.1) | 91.2 (4.6)
Statistical Analysis 1: Comparison: Glycine vs Placebo; Test type: Superiority or Other; p < 0.01, t-test, 1 sided; [statistical method as in outcome 1, analysis 1]

10. Secondary Outcome: Changes in Other Spirometric Variables
Description: as for outcome 8
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: Percentage of baseline
Arm/Group | Glycine | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of baseline
  Forced vital capacity (FVC) | 104.1 (4.1) | 100.6 (9.8)
  Forced expiratory flow at 75%FVC (FEF75) | 111.8 (11.7) | 108.9 (15.8)
Statistical Analysis 1: Comparison: Glycine vs Placebo; Test type: Superiority or Other; p > 0.05, t-test, 1 sided; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Weeks 4 and 8 of each study arm.
Groups:
- Glycine: Patients received a daily oral supplement of glycine at a dose of 0.5 g/kg divided in three doses during 8 weeks, dissolved in any liquid.
- Placebo: Patients received a daily oral supplement of sugar glass at a dose of 0.5 g/kg divided in three doses during 8 weeks, dissolved in any liquid.
Arm/Group | Glycine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No